CLINICAL TRIAL: NCT04789772
Title: Positive Effects of Laser Acupuncture in Methamphetamine Users Undergoing Group Cognitive Behavioral Therapy: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare (Ambiguous)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201800431A3
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Substance Abuse
Keywords: Substance abuse; Methamphetamine addiction; Laser acupuncture
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Because of uncertainty of effectiveness of laser acupuncture and drop out rate of MA users, investigators make an observational single group of pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser acupuncture group (Experimental): Laser acupuncture group receive laser acupuncture treatment with cognitive behavioral therapy.
  Interventions: Device: Laser acupuncture

INTERVENTIONS:
Device: Laser acupuncture — The interventional group receive laser acupuncture applied on acupoints of PC6 (Neiguan), HT7 (Shenmen), LI4 (Hegu), ST36 (Zusanli), SP6 (Sanyinjiao), and LR3 (Taichong).

SUMMARY:
Methamphetamine (MA) addiction has become a crucial public health issue due to its adverse effects. Acupuncture has been used for drug detoxification for many years. However, some disadvantages are not be suitable for MA users. The advantages of laser acupuncture includes safety, painless, less time consuming and higher acceptability without current investigation. Therefore, investigators arrange this study to evaluate the efficacy of laser acupuncture combined with golden treatment of cognitive group therapy.

DETAILED DESCRIPTION:
Methamphetamine (MA) addiction has become a crucial public health concern because of its adverse consequences to individuals and the society. Manual or auricular acupuncture have been applied in opioid dependence treatment for a long time. Electroacupuncture may also alleviate the symptoms of MA addiction such as psychosis, anxiety, and depression during abstinence. However, several comorbidities are associated with MA use, such as blood-borne infections, decreased the willingness of physicians to perform. The advantages of laser acupuncture (LA) include its safety, painlessness, limited time use, and higher acceptability, making it suitable for treatment of drug users. To investigate the clinical efficacy of laser acupuncture combined with group cognitive behavioral therapy for MA addiction treatment. MA users who participated in group cognitive behavioral therapy and met the inclusion criteria were referred from psychiatrists to participate. The participants received laser acupuncture treatment once a week for 2 months (total eight treatments) on selected acupoints (PC6, HT7, LI4, ST36, SP6, and LR3). Laboratory assessment included urinalysis for MA and liver function tests aspartate aminotransferase, alanine aminotransferase, and γ-glutamyltransferase (AST, ALT, and r-GT), whereas the objective assessment included visual analog scale (VAS) for MA craving and refusal and Pittsburgh sleep quality index (PSQI), Beck Anxiety Inventory (BAI), and Beck Depression Inventory (BDI) questionnaires. All data were collected before and at 1 and 2 months after treatment. Cognitive behavioral therapy completion rate and rate of relapse to MA use were also determined.

ELIGIBILITY:
Inclusion Criteria:

* subject must be aged ≥20 years, with full understanding of the content of the study and who signed a consent form
* subject must be diagnosed as MA use disorder by a psychiatrist according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
* subject must participate in cognitive behavioral therapy

Exclusion Criteria:

* subject received manual acupuncture or LA treatment in the preceding month
* subject had cancer, stroke, myocardial infarction, or major trauma
* subject demonstrated obvious suicide intention
* subject were pregnant
* subject were HIV-positive

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Change of Aspartate aminotransferase (AST) | change from baseline AST at 4 weeks and 8 weeks post-treatment
  To detect liver damage.
Change of Alanine aminotransferase (ALT) | change from baseline ALT at 4 weeks and 8 weeks post-treatment
  To detect liver damage.
Change of γ-glutamyltransferase (γ-GT) | change from baseline γ-GT at 4 weeks and 8 weeks post-treatment
  To detect liver damage.
Change of Amphetamine confirm test | change from baseline Amphetamine at 4 weeks and 8 weeks post-treatment
  To confirm drug exposure involving amphetamines.

SECONDARY OUTCOMES:
Change of Visual analog scale (VAS) | change from baseline VAS at 4 weeks and 8 weeks post-treatment
  Evaluation of MA craving and refusal from 0 to 10.
Change of Pittsburgh sleep quality index (PSQI) | change from baseline PSQI at 4 weeks and 8 weeks post-treatment
  Evaluation of sleep quality.
Change of Beck Anxiety Inventory (BAI) | change from baseline BAI at 4 weeks and 8 weeks post-treatment
  Evaluation the degree of anxiety.
Change of Beck Depression Inventory (BDI) | change from baseline BDI at 4 weeks and 8 weeks post-treatment
  Evaluation the degree of depression.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Center for traditional chinese medicine, Chang Gung Memorial Hospital, Guishan Dist, Taoyuan County
  - TSE-HUNG HUANG MD PhD, Keelung